CLINICAL TRIAL: NCT04974060
Title: Treatment of Spontaneous Hyperventilation in Severe Traumatic Brain Injury Patients: The Efficiency and Safety of Remifentanil Infusion and Its Impact on Cerebral Blood Flow
Brief Title: Treatment of Spontaneous Hyperventilation With Remifentanil in Traumatic Brain Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-002
Record Dates: First submitted 2021-04-08; First posted 2021-07-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hyperventilation; Traumatic Brain Injury
Keywords: Spontaneous Hyperventilation; Severe Traumatic Brain Injury; Cerebral Blood Flow; Remifentanil; Partial pressure of carbon dioxide
MeSH Terms: conditions — Hyperventilation; Brain Injuries, Traumatic | interventions — Remifentanil; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remifentanil intervention (Experimental): After the satisfactory analgesia and sedation, remifentanil will continuously infuse an escalating dose in the sequence of 0.02, 0.04, 0.06, and 0.08 μg/kg/min, each dose infusion lasting at least 30 minutes.
  Interventions: Drug: Remifentanil Injection

INTERVENTIONS:
Drug: Remifentanil Injection — Dilute 2mg Remifentanil with normal saline to 50 ml (40ug/ml) and continuously intravenous infused at the doses of 0.02, 0.04, 0.06, and 0.08 μg/kg/min for each lasting 30 minutes.
  Other Names: remifentanil hydrochloride for injection

SUMMARY:
Spontaneous hyperventilation is common in severe traumatic brain injury patients and correlates closely with poor outcomes. How to treat this pathological condition remain unsolved. Remifentanil is a frequently used short-acting opioid, has the potent side-effect of dose-dependent respiratory inhibition. Specifically, it prolongs the expiratory time only and does not influence the respiratory drive. Among the safety range, the investigators will determine an ideal dose of remifentanil to maintain PaCO2 between 35 to 45 mmHg. The investigators will monitor the cerebral blood flow of the middle cerebral artery and the internal carotid artery to validate cerebral perfusion improvement.

DETAILED DESCRIPTION:
Severe Traumatic Brain Injury (sTBI) is a devastating disease with high hospital mortality and disability worldwide. For neurocritical care physicians, avoiding secondary brain injury remains the cornerstone of treatment in treating sTBI patients.

Carbon dioxide is a potent cerebral vascular modulator. By decreasing the arterial partial pressure of carbon dioxide (PaCO2), hyperventilation could induce cerebral vasoconstriction and decrease cerebral blood flow (CBF), which further reduces cerebral blood volume and lowering intracranial pressure. Traditionally, intentional hyperventilation was used to control intracranial hypertension in sTBI patients for decades. However, evidences have shown that the decreased cerebral blood flow may aggravate brain ischemia and worse neural function. The most recent guidelines do not recommend prophylactic use of induced hyperventilation in sTBI patients anymore.

However, the latest research revealed a high prevalence of spontaneous hyperventilation (SHV) in sTBI patients, accompanied by prolonged sedation and analgesia, increased hospital mortality, and long-term adverse clinical outcomes. Although many modalities are available, there is still no consensus on the practical and feasible treatment for SHV in clinical practice.

As one of the most commonly used short-acting analgesic drugs, remifentanil has the characteristic of dose-depended respiratory rate inhibition by prolonging expiratory time, meanwhile preserve the respiratory drive. Among the effective dose range, the continuous infusion of remifentanil does not interfere the cerebral hemodynamics. The investigators hypothesize that SHV could be corrected with remifentanil infusion and anticipate increasing cerebral blood flow and improving the sTBI patients' outcomes.

This exploratory physiological study will titrate the respiratory rate with continuous remifentanil infusion in the sTBI patient with SHV, aiming to maintain the ideal PaCO2 range of 35-45 mmHg. Specifically, after the satisfactory analgesia and sedation achieved with butorphanol and midazolam/propofol, escalating remifentanil doses (0.02, 0.04, 0.06, and 0.08 ug/kg/min) will be tested in sequence from the baseline.

The parameters of vital signs, blood gas analysis, ventilator monitored variables such as tidal volume, minute ventilation, end-tidal carbon dioxide will be collected at the stable period after 30 minutes of drug infusion. Transcranial doppler also will be performed at the same time to evaluate the change of velocity of the middle cerebral artery and internal carotid artery. An efficient and safe dose range will be determined, meanwhile preserve the stability of neural function and hemodynamic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe TBI (3 < glasgow coma scale (GCS) ≤ 8)
* Hyperventilation (PaCO2 < 35 mmHg and pondus hydrogenii (pH) > 7.45)
* Presence of an endotracheal tube
* Assisted ventilation mode (CPAP/PSV)

Exclusion Criteria:

* Induced/iatrogenic hyperventilation
* No informed consent was signed
* Transcranial doppler sonography (TCD) data collection cannot be completed due to anatomical structure
* Severe multiple organ failure, persistent high fever, massive thoraco-peritoneal effusion
* Medical history of major craniocerebral injury and chronic obstructive pulmonary disease (COPD)
* Conformed or Suspected history of opioid-related adverse reactions
* Withdraw from the study due to the change of patient's condition and other methods of treatment and intervention are needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Explore the effective and safe dose of remifentanil to correct spontaneous hyperventilation in patients with severe traumatic brain injury | Baseline and 30 minutes following each infusion rate adjustment (0.02, 0.04, 0.06, and 0.08 μg/kg/min)
  The differences of partial pressure of carbon dioxide (PaCO2; mmHg) between the respective points (baseline and 30 minutes following each infusion rate adjustment of remifentanil) were recorded to determine the change of PaCO2 (mmHg).

SECONDARY OUTCOMES:
To explore the effect of remifentanil on the cerebral blood flow in patients with severe traumatic brain injury at the different dose of remifentanil | Baseline and 30 minutes following each infusion rate adjustment (0.02, 0.04, 0.06, and 0.08 μg/kg/min)
  Bilateral mean cerebral blood velocity changes of middle cerebral artery and internal carotid artery between baseline and 30 minutes following each infusion rate adjustment of remifentanil were recorded to determine the change of cerebral blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Intensive Care Unit, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Intensive Care Unit, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No